CLINICAL TRIAL: NCT03193034
Title: Multi-Center Clinical Evaluation of the ATTUNE® Cementless Rotating Platform Total Knee Arthroplasty in the Japanese Patient Population
Brief Title: DSJ-2016-07 ATTUNE® Cementless CR RP Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Collaborators: Johnson & Johnson K.K. Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSJ-2016-07
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty; replacement; Knee; function; radiographic; survivorship
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Masking Description: An independent radiographic reviewer will be assessing all radiographs from the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATTUNE Cementless RP TKA (Experimental): Subjects will receive a cementless, rotating platform total knee arthroplasty.
  Interventions: Device: Cementless Total Knee Arthroplasty

INTERVENTIONS:
Device: Cementless Total Knee Arthroplasty — Patients will undergo a primary total knee replacement using the configuration of the ATTUNE Cementless knee (CR RP)

SUMMARY:
The primary objective is to investigate the change from pre-operative baseline to two year postoperative functional performance improvement for the ATTUNE® primary, cementless TKA RP system as measured with the KOOS questionnaire (KOOS-ADL sub-score) in the Japanese patient population.

DETAILED DESCRIPTION:
* Evaluate change from preoperative baseline in post-operative outcomes using additional patient reported measures at 2 years: PKIP (overall and sub-scores), KOOS (overall and sub-scores), AKS and EQ-5D-3L.
* Evaluate change from preoperative baseline in pain and satisfaction over time as measured using a modified VAS Pain Score (discrete numbers rather than a continual scale) at 2yr.
* Evaluate type and frequency of Adverse Events
* Evaluate survivorship of the ATTUNE® Primary Cementless TKA system for the CR RP configurations using Kaplan-Meier survival analysis at 1 and 2yrs.
* Evaluate primary, cementless ATTUNE® TKA fixation through zonal radiographic analysis of the bone-implant interface at 6wk, 1yr, and 2yrs after surgery.
* Evaluate any changes in anatomic tibiofemoral, femoral component and tibial component alignment at 2 years compared to the first postoperative radiographs.
* Radiographically characterize the postoperative ATTUNE patellar component alignment and positioning in Japanese population.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and between the ages of 22 and 80 years at the time of surgery, inclusive.
* Subject was diagnosed with NIDJD.
* Subject, in the opinion of the Investigator, is a suitable candidate for cementless primary TKA using the devices described in this CIP with either resurfaced or non-resurfaced patellae.

Subject that is willing to give voluntary, written informed consent to participate in this clinical investigation and authorize the transfer of his/her information to the Sponsor .

* Subject is currently not bedridden
* Subject, in the opinion of the Investigator, is able to understand this clinical investigation and is willing and able to perform all study procedures and follow-up visits and co-operate with investigational procedures.
* Subject is able to read, and comprehend the Informed Consent Document as well as complete the required PROs in Japanese.

Exclusion Criteria:

* The Subject is a woman who is pregnant or lactating. -Contralateral knee has already been enrolled in this study
* Subject had a contralateral amputation.
* Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or primary TKA in affected knee.
* Subject is currently diagnosed with radicular pain from the spine that radiates into the limb to receive TKA.
* Subject has participated in a clinical investig ation with an investigational product (drug or device) in the last three (3) months.
* Subject is currently involved in any personal injury litigation, medical-legal or Worker's Acc ident Insurance claims (similar to Workers Compensation in USA).
* Subject, in the opinion of the Investigator, is a drug or alcohol abuser (in the last 5 years) or has a psychological disorder that could affect their ability to complete patient reported question naires or be compliant with follow-up requirements.
* Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
* Subject has a significant neurological or musculoskeletal disorder(s) or disease that may adversely affect gait or weight bearing (e.g., muscular dystrophy, multiple sclerosis, Charcot disease).
* Subject is suffering from inflammatory arthritis (e.g., rheumatoid arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, etc.).
* Subject has a medical condition with less than two (2) years life expectancy.
* Uncontrolled gout

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Patient-reported Outcome:Knee Injury and Osteoarthritis Outcome Score Activities of Daily Living (KOOS ADL) | Minimum 2 years (670-912 days after surgery)
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient self-administered questionnaire that consists of 42 questions and include the WOMAC Osteoarthritis index. The KOOS consists of 5 subscales: pain, other symptoms, activities of daily living (ADL), sport and recreational function and knee related quality of life. Each question has 5 Likert-like response options. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.

SECONDARY OUTCOMES:
Patient-reported Outcome: Pre-surgical/Post-surgical Patient's Knee Implant Performance (PKIP) | Minimum 2 years (670-912 days after surgery)
  The Pre Surgical and/or Post-surgical Patient's Knee Implant Performance (PKIP) questionnaire is a patient self-administered questionnaire that consists of 25 questions relating to the patient's awareness of their knee. Questions include the patient's self-confidence about the current status of their knee performance, stability, and overall satisfaction. Each question has a 5, 6 or 10 Likert- like response option.
Patient-reported Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) | Minimum 2 years (670-912 days after surgery)
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient self-administered questionnaire that consists of 42 questions and include the WOMAC Osteoarthritis index. The KOOS consists of 5 subscales: pain, other symptoms, activities of daily living (ADL), sport and recreational function and knee related quality of life. Each question has 5 Likert-like response options. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Combination of Patient-reported and Clinical-reported Outcome: Knee Society 2011 | Minimum 2 years (670-912 days after surgery)
  The Knee Society Score is a self-administered questionnaire. The subject completes questions regarding: Symptoms (3 questions), Patient Satisfaction (5 questions), Patient Expectations (3 questions), Functional Activities (5 questions), Standard Activities (6 questions), Advanced Activities (5 questions), and Discretionary Knee Activities ( 4 questions). The surgeon completes questions regarding objective knee indicators. Likert responses are used, typically with five response options.
Patient Reported Outcome: EuroQol 5D 3L questionnaire (EQ-5D-3L) | Minimum 2 years (670-912 days after surgery)
  EuroQol 5D 3L questionnaire is a standardized instrument for use as a measure of health outcome that is designed for completion by the subject.
Modified VAS Pain Score: Pain and Satisfaction | Minimum 2 years (670-912 days after surgery)
  VAS Pain Score is a standardized instrument for use as a measure of pain and satisfaction that is designed for completion by the subject. This modified version has scores that are discrete numbers rather than a continual scale
Type and Frequency of Adverse Events (AEs) for all enrolled subjects | Pre-op (-180 to -1 days before surgery), 6 weeks (1-303 days after surgery), minimum 1 year (304-669 days after surgery), minimum 2 years (670-912 days after surgery)
  All Serious AEs must be reported to Sponsor. All device-related or procedure-related adverse events must be reported to Sponsor.
Survivorship | Minimum 1 year (304-669 days after surgery), minimum 2 years (670-912 days after surgery)
  Kaplan-Meier survival analysis will be used to calculate the survivorship of configuration (CR RP)
Implant fixation: Radiographic assessment of bone-implant interface performance | 6 weeks (1-303 days after surgery), minimum 1 year (304-669 days after surgery), minimum 2 years (670-912 days after surgery)
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Evaluate changes in femoral component and tibial component alignment | Minimum 2 years (670-912 days after surgery)
  Radiographic success is defined as: absence of progressive radiolucent lines greater than or equal to 2mm in any one zone; absence of lytic lesions in any zone; absence of individual component position change >3degrees in any plane.
Radiographically characterize the postoperative ATTUNE patellar component alignment and positioning in Japanese population. | Minimum 1 year (304-669 days after surgery)
  Evaluate the tilt angle and translational position of the patellar component relative to the trochlear groove.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Cosgrove, Study Director — Sponsor GmbH
Locations (4):
- Japan (4):
  - Nagoya orthopedic Clinic, Kitanagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Kobe University Graduate School of Medicine, Kobe, Hyōgo
  - Osaka Rosai Hospital, Sakai, Osaka

IPD SHARING:
Plan to Share IPD: Undecided